CLINICAL TRIAL: NCT03192956
Title: Neuroskademarkörer Vid Dykarsjuka
Brief Title: Markers of Central Nervous System Injury in Decompression Sickness
Acronym: DCS NEURO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Anders Rosén, MD PhD, Sahlgrenska University Hospital
Other Study IDs: EPN 552-16
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Decompression Sickness
Keywords: Hyperbaric; Decompression sickness; Decompression injury; Inflammation; Central nervous injury; Hybervaric oxygen therapy
MeSH Terms: conditions — Decompression Sickness; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum. Plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No active intervention — No active intervention is performed

SUMMARY:
Research hypothesis

* There is a correlation between the quantity of fluid markers of CNS injury in blood and DCS.
* There is a correlation between quantity and kind of fluid markers of CNS injury in blood and both diving profile and severity of DCS.
* There is a correlation between the quantity of inflammatory markers in blood an DCS.

Objectives:

* Assess whether individuals suffering decompression sickness exhibit fluid markers of central nervous system injury.
* Evaluate the correlation between quantity and kind of fluid marker of CNS injury and clinical signs of neurological impairment.
* Evaluate the correlation between quantity and kind of fluid marker of CNS injury and clinical outcome after 3-6 months.
* Assess whether individuals suffering decompression sickness exhibit inflammatory markers in blood.

DETAILED DESCRIPTION:
Decompression sickness (DCS) is a risk associated with diving. Common symptoms are joint and limb pain, skin rash, ataxia, hemiplegia, visual disturbances, paresthesias, limb numbness, nystagmus and vertigo. Treatment consists of recompression in a hyperbaric chamber, commonly referred to as hyperbaric oxygen treatment (HBOT).

It has been thought since the last quarter of the 19th century that DCS is caused by bubble formation in the tissues when dissolved inert gas comes out of solution. It was long thought that decompression schedules that did not give rise to any gas bubbles in the body also averted DCS. However, with the advent of ultrasound Doppler technology in the 1970s it was found that intravascular gas bubbles could exist even after uneventful dives. Dives well within limits established by military and sports authorities have been shown to generate intravascular bubbles. Hence, additional pathophysiological factors have been sought.

There is evidence of endothelial dysfunction, coagulopathy and inflammatory activation after diving. Though, their role in the pathophysiology of DCS remains to be determined.

Studies have shown that fluid markers of CNS injury can be found in blood samples obtained from athletes practising ice-hockey, boxing and american football. There is reason to believe that fluid markers of CNS injury will be present in blood samples obtained from divers with DCS as well.

Study subjects will be recruited by the attending physician at the Hyperbaric chamber at SU/Omrade 2 after the patient has been given a diagnosis of decompression sickness. Prior to treatment in the hyperbaric chamber, 4 ml of blood will be drawn via a plastic intravenous catheter that is placed in an arm vein as part of normal, established care of injured divers in the Emergency Department (to provide intravenous fluid and medications). A second 4 ml sample will be obtained from the same catheter after the patient has completed treatment (the typical hyperbaric treatment for decompression sickness lasts ~5.5 hours). The study object will also provide information regarding his/her general health and the completed dive. All study data, including blood samples, will anonymized and provided with a study code.

When feasible, blood samples will be obtained 1 week and 3-6 months after HBOT. These samples will be handled the same as the two obtained on the day of injury.

ELIGIBILITY:
Inclusion Criteria:

* Presence of decompression sickness
* Signed informed consent

Exclusion Criteria:

* As this is a highly selected population there is no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research subjects are recruited, on voluntary basis, among divers with decompression sickness treated at the hyperbaric facility at Sahlgrenska Universuty Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical signs of central nervous system injury | 6 months
  E. g: Tau, NfL, GFAP, UCHL-1

SECONDARY OUTCOMES:
Inflammatory activity | 6 months
  E. g: VCAM-1, ICAM-1, Endothelin-1
Symptoms of decompression sickness | 24 hours
  Clinical diagnosis
Dive time | 1 hour
  Minutes
Dive depth | 1 hour
  Meters of seawater
Remaining symptoms of decompression sickness after 3-6 months | 6 months
  Clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Zetterberg, PhD, Study Director — Göteborg University
Locations (1):
- Gothenburg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No